CLINICAL TRIAL: NCT06874062
Title: Clinical and Radiographic Evaluation of the Success of Resin-Modified Calcium Silicate in Primary Tooth Pulpotomy
Brief Title: Evaluation of Primary Tooth Pulpotomy With Resin Modified Calcium Silicate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Rabia Yücel, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/257
Record Dates: First submitted 2025-03-03; First posted 2025-03-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Pulpotomy
Keywords: pulpotomy; mineral trioxide aggregate; resin-modified calcium silicate cement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NeoPutty MTA (Experimental): A ready-to-use putty-form Neoputty® MTA with a minimum piston length of 1.5 mm was placed on the pulp chamber floor using a sterile dental spatula. The material was adapted to the canal orifices with the aid of a cotton pellet that had been lightly moistened with sterile saline.
  Interventions: Procedure: Neoputty MTA Pulpotomy Treatment; Procedure: Stainless Steel Crown Application
- ProRoot MTA (Experimental): Using a sterile glass and spatula, an adequate amount of powder and liquid was mixed for approximately 1 minute until a homogeneous consistency was achieved, following the manufacturer's recommendations. The ProRoot® MTA, prepared to a putty-like consistency, was transferred to the pulp chamber using a sterile dental spatula and adapted to the canal orifices with the aid of a cotton pellet.
  Interventions: Procedure: ProRoot MTA Pulpotomy Treatment; Procedure: Stainless Steel Crown Application
- Theracal PT (Experimental): The TheraCal PT® package contains a 4 g tube and 10 single-use mixing tips. One of the disposable mixing tips was attached to the tube, and the material was mixed within the tip by pressing the plunger. The material was then directly applied to the pulp chamber. Adaptation of the material to the canal orifices was verified using a sterile cement applicator. Polymerization was performed for 10 seconds using a Woodpecker LED B (Guilin Woodpecker Medical Instrument Co., Ltd., China) curing light device, following the manufacturer's instructions.
  Interventions: Procedure: Theracal PT Pulpotomy Treatment; Procedure: Stainless Steel Crown Application

INTERVENTIONS:
Procedure: Neoputty MTA Pulpotomy Treatment — All caries were removed before entering the pulp chamber. Once all caries were removed, a carbide bur was used under copious water spray to expose the pulp chamber.Coronal pulp is removed with a round bur on a slow speed handpiece.
  Hemostasis was achieved by applying a cotton pellet moistened with sterile saline for no more than 5 minutes. After achieving hemostasis, Neoputty MTA was placed.
  Arms: NeoPutty MTA
Procedure: ProRoot MTA Pulpotomy Treatment — All caries were removed before entering the pulp chamber. Once all caries were removed, a carbide bur was used under copious water spray to expose the pulp chamber.Coronal pulp is removed with a round bur on a slow speed handpiece.
  Hemostasis was achieved by applying a cotton pellet moistened with sterile saline for no more than 5 minutes. After achieving hemostasis, ProRoot MTA was placed.
  Arms: ProRoot MTA
Procedure: Theracal PT Pulpotomy Treatment — All caries were removed before entering the pulp chamber. Once all caries were removed, a carbide bur was used under copious water spray to expose the pulp chamber.Coronal pulp is removed with a round bur on a slow speed handpiece.
  Hemostasis was achieved by applying a cotton pellet moistened with sterile saline for no more than 5 minutes. After achieving hemostasis, Theracal PT was placed.
  Arms: Theracal PT
Procedure: Stainless Steel Crown Application — After pulpotomy treatment, the pulpotomy material was covered using a capsule-form glass ionomer (EQUIA Forte®, GC, Tokyo, Japan). In the same session, preparation was performed for the placement of a stainless steel crown (SSC), and an appropriately sized SSC (3M ESPE, Seefeld, Germany) was selected based on visual estimation. After trial fitting on the tooth, the crown was cemented using a capsule-form glass ionomer (Riva, SDI Ltd., Victoria, Australia).

SUMMARY:
The goal of this clinical trial is to evaluate whether Theracal PT, a resin-modified calcium silicate-based material, can be successfully used in pulpotomy treatment for primary molar teeth. The efficacy of this material will be compared with MTA in its putty form (Neoputty) and powder-liquid form (ProRoot). The main questions this study aims to answer are: Is Theracal PT as effective as MTA, the gold standard for pulpotomy treatment? Is Neoputty MTA, which is easier to handle, more effective than ProRoot MTA? The study will include systemically healthy children aged 4 to 9 years with at least one primary molar requiring pulpotomy. Treated teeth will be evaluated clinically and radiographically at 3, 6, and 12 months.

DETAILED DESCRIPTION:
Tooth decay is a complex process of enamel demineralization and remineralization caused by organic acids produced by microorganisms in the dental plaque. When this balance shifts in favor of demineralization, caries formation occurs. Initially, decay begins with small surface roughness or subsurface demineralization, followed by cavitation and subsequent pulp involvement.

Tooth decay, one of the most common chronic diseases in childhood, negatively impacts the quality of life when left untreated, leading to problems such as pain, abscess formation, tooth loss, nutritional deficiencies, and speech disorders. To prevent early loss of primary teeth and maintain the health of the oral and surrounding tissues, restorative or endodontic treatments are applied. Treatment methods for deep dentin caries in primary teeth include indirect pulp capping, direct pulp capping, and amputation, with amputation being the most commonly used vital pulp therapy. Amputation is indicated when the pulp is either healthy or reversibly damaged and shows no signs of pulp degeneration, and the pulp becomes exposed during caries removal due to decay or mechanical causes. The goal of treatment is to preserve the vitality of the radicular pulp, control pain and inflammation, and maintain the tooth until its physiological exfoliation time. The selection of appropriate materials and techniques for amputation therapy is of critical importance. Although several studies have investigated the success of amputation materials and techniques, the ideal amputation material has not yet been defined. The ideal material and technique should be bactericidal, harmless to the pulp and surrounding tissues, support the healing of the root pulp, and contribute to the preservation of remaining tissues without affecting physiological root resorption. Additionally, factors such as cost and ease of application should also be considered in material selection. Therefore, efforts to identify the ideal amputation material continue.

The aim of this study is to evaluate the clinical and radiographic success of Theracal PT®, ProRoot® MTA, and Neoputty® MTA, and to examine the relationship between these outcomes and factors such as age, gender, the position of the tooth in the arch, and the presence of provoked pain prior to treatment.

The following hypotheses were proposed in our study:

Hypothesis 1: There is no difference in the 12-month clinical and radiographic success rates of primary tooth amputation treatments performed using Neoputty® MTA, ProRoot® MTA, and Theracal PT®.

Hypothesis 2: The 12-month clinical and radiographic success of amputation treatments performed using Neoputty® MTA, ProRoot® MTA, and Theracal PT® is not influenced by age, gender, the position of the tooth in the arch, or the presence of provoked pain prior to treatment.

This study was conducted in accordance with the Ataturk University Faculty of Medicine Ethics Committee approval (Date: 30.03.2023/ Session no:02/ Decision no:04) and guidelines of the Helsinki Declaration. The study was supported by the Scientific Research Projects Coordination Unit of Atatürk University under project number TDH-2023-13045. In this study, the teeth to be treated were randomly assigned using stratified randomization, ensuring an equal number of teeth in each study group. The research design was based on a parallel groups model. When multiple teeth from the same patient participated in the study, randomization was also applied for the other materials to be used. Patient selection, examination, treatment, and follow-up processes were carried out by a single researcher undergoing specialty training in the Department of Pediatric Dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Deep dentin caries,
* Lamina dura and periodontal interval can be observed normally,
* 2/3 of the root length is present,
* The permanent tooth germ below is present and its position is normal,
* If there is a history of provoked pain (the type of pain that goes away when the stimulus is removed),
* If there is a history of pain (short-term provoked pain, the pain goes away when the stimulus is removed,
* Teeth with mechanical perforation larger than a needle tip in the perforation area or perforated with caries,
* Teeth with light-colored bleeding and easily controlled within 3-5 minutes,
* Teeth that can be restored with PÇK were included in the study

Exclusion Criteria:

* Lesions in the inter-root and periapical region,
* Pathological external or internal root resorption,
* Canal calcification,
* Deformities such as taurodontism,
* Spontaneous pain or night pain,
* Structural anomalies,
* Abscess, swelling or fistula,
* Pathological mobility,
* Sensitivity to palpation and percussion,
* Infraocclusion,
* Dark, intense bleeding in the canal orifices

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Clinical Success | 1 Month - 1 Year
  No spontaneous, provoked (developing due to a stimulus) or night pain complaints.
  No sensitivity to percussion or palpation. No pathological mobility in the tooth. No abscess or fistula in the tooth. If any of these findings are detected, the treatment is considered clinically unsuccessful.
Radiographic Success | 3 Month - 1 Year
  No internal or external root resorption. No periapical or inter-root lesion. No widening of the periodontal space. If any of these findings are detected, the treatment is considered radiographically unsuccessful.

SECONDARY OUTCOMES:
The Impact of Patient's Age on 12-Month Radiographic Success of Treatment. | From treatment to the end of 12 months
  The patient's age was compared with the radiographic success parameters at 12 months. Radiographic success parameters:
  No internal or external root resorption. No periapical or inter-root lesion. No widening of the periodontal space.
The Impact of Patient's Gender on 12-Month Radiographic Success of Treatment. | From treatment to the end of 12 months
  The patient's gender was compared with the radiographic success parameters at 12 months. Radiographic success parameters:
  No internal or external root resorption. No periapical or inter-root lesion. No widening of the periodontal space.
The Impact of Tooth Position in the Dental Arch on the 12-Month Radiographic Success of Treatment | From treatment to the end of 12 months
  The tooth position in the dental arch was compared with the radiographic success parameters at 12 months. Radiographic success parameters:
  No internal or external root resorption. No periapical or inter-root lesion. No widening of the periodontal space.
The Impact of Pre-Treatment Provoked Pain on the 12-Month Radiographic Success of Treatment. | From treatment to the end of 12 months
  The presence of provoked pain before treatment in the patient was compared with radiographic success parameters at the 12th month. Radiographic success parameters:
  No internal or external root resorption. No periapical or inter-root lesion. No widening of the periodontal space.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Şengül, Phd, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordell S, Kratunova E, Marion I, Alrayyes S, Alapati SB. A Randomized Controlled Trial Comparing the Success of Mineral Trioxide Aggregate and Ferric Sulfate as Pulpotomy Medicaments for Primary Molars. J Dent Child (Chic). 2021 May 15;88(2):120-128. PMID 34321144
- [Background] Waterhouse P. Are different pulp treatment techniques and associated medicaments effective for the treatment of extensive decay in primary teeth? Evid Based Dent. 2021 Jan;22(1):12-13. doi: 10.1038/s41432-021-0162-6. PMID 33772121
- [Background] Celik B, Atac AS, Cehreli ZC, Uysal S. A randomized trial of mineral trioxide aggregate cements in primary tooth pulpotomies. J Dent Child (Chic). 2013 Sep-Dec;80(3):126-32. PMID 24351693
- [Background] Wassel M, Hamdy D, Elghazawy R. Evaluation of four vital pulp therapies for primary molars using a dual-cured tricalcium silicate (TheraCal PT): one-year results of a non-randomized clinical trial. J Clin Pediatr Dent. 2023 Mar;47(2):10-22. doi: 10.22514/jocpd.2023.004. Epub 2023 Mar 3. PMID 36890738